CLINICAL TRIAL: NCT04508673
Title: Comparative Study of Human Growth Hormone Measurements: Impact on Clinical Interpretation
Brief Title: Impact of GH Measurements on GHD Diagnosis
Status: Completed | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL20_0449
Record Dates: First submitted 2020-08-07; First posted 2020-08-11 (Actual); Last update posted 2020-08-17 (Actual); Status verified 2020-08

CONDITIONS: Growth Hormone Deficiency
Keywords: growth hormone deficiency; immunoanalysis; hGH provocation test; diagnosis
MeSH Terms: conditions — Dwarfism, Pituitary; Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — serum
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: GH provocation tst — All patients underwent insulin-induced hypoglycaemia stimulation test also called insulin tolerance test (ITT), considered the 'gold standard' test for GHD diagnosis. Following insulin administration by venipuncture (1UI/mL), levels of hGH and glucose were monitored on serum and fluoride tube plasma, respectively, at intervals of 0, 30, 45, 60 and 90 minutes (T0, T30, T45, T60 and T90).
  Other Names: reliquens of serum samples from GH provocation test

SUMMARY:
Human growth hormone (hGH) provocation test is an essential tool to assess growth hormone deficiency in children and young adults. It is important to have a robust and reliable method to determine the hGH peak of stimulation. This work aimed to compare three common automated immunoassays for hGH measurements and to assess whether there are still result-related differences influencing clinical decision.

DETAILED DESCRIPTION:
The investigators analysed GH provocative test of 41 young patients (median age: 12 years) from Pediatric Department of Montpellier Hospital, (26 boys and 15 girls), admitted for follow-up or for suspicion of growth hormone deficiency. Serum GH of peak concentrations were compared using three automated immunoanalyses : COBAS 8000 e602 (ROCHE Diagnostics), IDS-iSYS (IDS immunodiagnostic systems) and Liaison XL (Diasorin S.A.).

ELIGIBILITY:
Inclusion criteria:

* Age<18 years, admitted for suspicion (short stature or growth retardation) or follow-up of GHD in pre-and pubertal age
* patients undergoing insulin-induced hypoglycaemia stimulation test also called insulin tolerance test (ITT)
* Exclusion criteria:
* Age > 18 years
* Patients undergoing different provocation tests

Ages: 9 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: From April to November 2019, forty-one young patients (26 boys and 15 girls) from the Paediatric Department of Montpellier Hospital were included in this study. They were mainly admitted for suspicion (short stature or growth retardation) or follow-up of GHD in pre-and pubertal age (median age= 12).
Sampling Method: Probability Sample
Enrollment: 41 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2019-11-01 (Actual); Study Completion 2019-11-25 (Actual)

PRIMARY OUTCOMES:
Comparative study of human growth hormone measurements | 1 day
  Comparative study of human growth hormone measurements by using three different automated immunoassays

SECONDARY OUTCOMES:
Stratification of patients based on GH peak secretion | 1 day
  Stratification of patients based on GH peak secretion

CONTACTS AND LOCATIONS:
Overall Officials: Manuela Lotierzo, PhD, Principal Investigator — UH MONTPELLIER
Locations (1):
- Uhmontpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided
NC

REFERENCES:
- [Derived] Lotierzo M, Olaru-Soare F, Dupuy AM, Plawecki M, Paris F, Cristol JP. Comparative study of human growth hormone measurements: impact on clinical interpretation. Clin Chem Lab Med. 2021 Dec 2;60(2):191-197. doi: 10.1515/cclm-2021-1109. Print 2022 Jan 27. PMID 34850616